CLINICAL TRIAL: NCT02176824
Title: Adjunct Total Sleep Deprivation, Sleep Phase Advance, and White Light Therapy Vs. Partial Sleep Deprivation, Sleep Phase Delay, and Amber Light Therapy as Adjunctive Treatments in Acutely Suicidal and Depressed Inpatients.
Brief Title: Chronotherapy Randomized Controlled Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Chronotherapy RCT
Record Dates: First submitted 2014-06-24; First posted 2014-06-27 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Major Depressive Disorder; Bipolar Depression; Suicidal Ideation
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Suicidal Ideation | interventions — Ultraviolet Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Triple Chronotherapy (Experimental): Total Sleep Deprivation, Sleep phase advance, and Bright Light Therapy. Carex Health Brands Day-Light Classic 10,000 Lux
  Interventions: Behavioral: Total Sleep deprivation, Sleep Phase Advance, and Bright Light Therapy
- Sham Triple Chronotherapy (Sham Comparator): Total sleep deprivation, Three day fixed wake schedule, and sham light therapy.
  Interventions: Behavioral: Partial Sleep deprivation, Sleep Phase Delay, and Low amber light.
- Treatment As Usual (Active Comparator): Normal inpatient care including pharmacotherapy, psychotherapy, milieu therapy, and social work interventions.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Total Sleep deprivation, Sleep Phase Advance, and Bright Light Therapy — Sleep deprivation, Sleep phase advance, and Bright light therapy
  Arms: Triple Chronotherapy
Behavioral: Partial Sleep deprivation, Sleep Phase Delay, and Low amber light.
  Other Names: Carex Health Brands Day-Light Classic 10,000 LUX with custom amber filter from lowbluelights.com
  Arms: Sham Triple Chronotherapy
Other: Treatment as usual
  Arms: Treatment As Usual

SUMMARY:
Chronotherapy is a term that describes therapeutic alterations of sleep wake cycles. Different variations of sleep deprivation, set sleep wake schedules, and types of light therapy have demonstrated efficacy in rapidly treating depression, and suicidal thinking. This study seeks to explore the effect of two different chronotherapuetic protocols on acutely depressed and suicidal inpatients admitted to the Medical University of South Carolina

DETAILED DESCRIPTION:
There is a consistently reported, rapid antidepressant response to a single night of total sleep deprivation in both unipolar, and bipolar depression. The clinical utility of this technique has been limited however, because responders have typically relapsed rapidly following recovery sleep. The addition of pharmacotherapy, sleep phase advance (a shift to an earlier sleep schedule with normalization over three days), and bright light therapy to sleep deprivation have each demonstrated efficacy in preventing relapse into depression. Combined total sleep deprivation, sleep phase advance, and bright light therapy, dubbed Triple Chronotherapy along with concomitant pharmacotherapy has demonstrated a rapid improvement in depressive symptoms that has remained durable for as long as 9 weeks post intervention. If the early, encouraging results of Triple Chronotherapy hold up to further study, the technique represents a near ideal inpatient treatment, as it is inexpensive, relatively easy to carry out, and has minimal side effects.

Despite encouraging early results, only one published report has attempted to use triple chronotherapy in suicidal patients, and in that trial only bipolar depressed patients were included, and one single variation of chronotherapy was tested (Three nights of sleep deprivation every other night with three light therapy sessions, combined with lithium). The lack of data in acutely suicidal patients significantly limits the utility of this intervention in the United States, where few non-suicidal patients are admitted. Published trials to this point have also excluded those with comorbid illness, which also limits the clinical usefulness of this intervention to a minority of patients. Furthermore there are sparse randomized adequately controlled trials, and still limited durability data on the technique.

We recently explored the tolerability and feasibility of the technique on acutely depressed and suicidal inpatients admitted to our inpatient unit with encouraging results. We subsequently propose to further explore the utility of this technique by piloting its effect compared to an active sham condition to determine if further study is indicated. Should further study be warranted, we hope to use the collected pilot data to determine the necessary number of participants to detect an effect.

ELIGIBILITY:
Inclusion Criteria:

* A current episode of non-psychotic major depression
* Currently hospitalized
* Age greater than 18
* If bipolar illness, must not be a mixed state, and must be on a therapeutic dose of a mood stabilizer

Exclusion Criteria:

* Urine drug screen positive for cocaine, or current alcohol/dependence that requires detox
* current psychosis
* Panic Disorder
* Severe Borderline Personality Disorder
* A history of seizures, uncontrolled severe headaches, stroke, or other neurologic illness that produces either gait abnormalities or lowered seizure threshold
* Medical illness that would make wake therapy intolerable
* Cataracts, glaucoma, or other intrinsic eye condition
* Currently taking light sensitizing medications
* Current pregnancy
* Mental retardation or dementia
* Untreated sleep disorder such as Obstructive Sleep Apnea(OSA), narcolepsy, or periodic limb movement disorder(PLMD) that results in excessive sleepiness
* Currently receiving electroconvulsive therapy (ECT)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-06-01; Primary Completion 2016-04-07 (Actual); Study Completion 2016-04-07 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | Day prior to total sleep deprivation, and then again over the next 4 consecutive days. There will then be a continuation phase where data will be collected at one week, two weeks, 4 weeks, and 8 weeks.
  Change in scores from Pre and Post Hamilton Depression scores
Columbia Suicide Severity Rating Scale | Day prior to total sleep deprivation, and then again over the next 4 consecutive days. There will then be a continuation phase where data will be collected at one week, two weeks, 4 weeks, and 8 weeks.
  Change in score of Columbia Suicide Severity Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Sahlem, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States